CLINICAL TRIAL: NCT01027117
Title: A Randomised, Open-Label 3-Way Crossover Study To Investigate The Relative Bioavailability Of The Crushed Revatio 20 Mg Tablet Mixed With Apple Sauce, The Extemporaneously Prepared Suspension (EP), And The Intact Revatio 20 Mg Tablet In Healthy Volunteers Under Fasting Conditions
Brief Title: A Relative Bioavailability Study of Revatio for the Crushed Tablets, Extemporaneously Prepared Formulation, and the Intact Tablets at 20 mg Dose in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A1481275
Record Dates: First submitted 2009-09-29; First posted 2009-12-07 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: Bioavailability; Revatio; Healthy Volunteers
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Active Comparator): Revatio 20 mg intact tablet. This is the reference treatment arm.
  Interventions: Drug: Revatio
- Treatment B (Experimental): Treatment B: Revatio 20 mg crushed tablet mixed with apple sauce.
  Interventions: Drug: Revatio
- Treatment C (Experimental): Treatment C: Revatio 20 mg extemporaneously prepared suspension (EP).
  Interventions: Drug: Revatio

INTERVENTIONS:
Drug: Revatio — Three treatments as described in study design, single dose, three way crossover. The treatment duration will be minimum 3 days for each subject.
  Arms: Treatment A
Drug: Revatio — Three treatments as described in study design, single dose, three way crossover. The treatment duration will be minimum 3 days for each subject.
  Arms: Treatment B
Drug: Revatio — Three treatments as described in study design, single dose, three way crossover. The treatment duration will be minimum 3 days for each subject.
  Arms: Treatment C

SUMMARY:
This will be a randomized, open-label, 3-treatment, 3-period, crossover, single-dose study in healthy subjects. Eighteen (18) subjects will complete the study; dropouts may be replaced at the discretion of the sponsor. Three treatments are:

Treatment A: Revatio 20 mg intact tablet. Treatment B: Revatio 20 mg crushed tablet mixed with apple sauce. Treatment C: Revatio 20 mg extemporaneously prepared suspension (EP). Blood samples for the analysis of sildenafil in plasma will be obtained pre-dose and up to 14 hours post dose in each period. Tolerability and safety will be assessed by reported adverse events during each study period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male/female subjects between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject or a legally acceptable representative.
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, ocular or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at Screening.
* History of febrile illness within 5 days prior to the first dose.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
AUClast | Within 14 hours post dose
Cmax | Within 14 hours post dose

SECONDARY OUTCOMES:
T1/2 | Within 14 hours post dose
AUCinf | Within 14 hours post dose
Tmax | Within 14 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium